CLINICAL TRIAL: NCT04731792
Title: Therapeutic Virtual Reality: Helps Reduce Anxiety and Pain During Bronchial Fibroscopies in Lung Transplant Patients.
Acronym: REVDOU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-A00658-31
Record Dates: First submitted 2021-01-21; First posted 2021-02-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Anxiety; Stress; Pain; Bronchial Fibroscopy; Pulmonary Transplantation
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality group (Experimental)
  Interventions: Other: Virtual Reality
- control group (No Intervention)

INTERVENTIONS:
Other: Virtual Reality — a bronchial fibroscopy with a virtual reality helmet
  Arms: Virtual Reality group

SUMMARY:
Marie Lannelongue Hospital is a hospital specialized in lung transplantation. Lung transplant patients require regular check-ups by bronchial fibroscopy. This examination is known to be anxious, stressful and sometimes painful. These patients take many medications (immunosuppressants, antibiotics....) that may interact with analgesic or anxiolytic drugs.

The objective is to propose to HML lung transplant patients a virtual reality solution containing visual and auditory 3D experiences to fight against anxiety and pain during repetitive and anxiogenic examinations such as bronchial fibroscopies.

Translated with www.DeepL.com/Translator (free version)

ELIGIBILITY:
Inclusion Criteria:

* Patient with a lung or cardio-pulmonary transplant
* Adults (age > 18 years old)
* Patient who give their informed consent for the protocol
* Patient requiring a bronchial fibroscopy and having already had at least one - bronchial fibroscopy without virtual reality

Exclusion Criteria:

- children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2021-01-14 (Actual); Primary Completion 2024-01-14 (Estimated); Study Completion 2024-02-14 (Estimated)

PRIMARY OUTCOMES:
Visual Analogic Scale (VAS) score from 0 (no anxiety) to 10 (terrified). | 1 day

SECONDARY OUTCOMES:
Evaluation of pain by a score on a numerical scale (EN) from 0 (no pain) to 10 (unbearable pain) | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Chirurgical Marie Lannelongue, Le Plessis-Robinson, France